CLINICAL TRIAL: NCT03741777
Title: Comparison of Residual Gastric Volume Between Children Who Drink Different Clear Oral Fluid Volume Before Undergoing Elective Esophago-gastro-duodenoscopy (EGD) Procedure
Brief Title: Comparison of Residual Gastric Volume Between Children Who Drink Different Clear Oral Fluid Volume
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Patcharee Sriswasdi, Attending staff, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00029632
Record Dates: First submitted 2018-08-29; First posted 2018-11-15 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Fasting; Gastric Emptying
Keywords: NPO time; Gastric content
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Intervention Model Description: The children included in this study will be randomly assigned into one of four groups by using randomization.org: Group 1 will consume 3 ml/kg of clear fluid by mouth at 2-hour period before surgical scheduled time, Group 2 will consume 5 ml/kg, Group 3 will consume 7 ml/kg, and Group 4 will consume 10 ml/kg.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3 ml/kg of clear oral fluid (Active Comparator): This group of patient will consume 3 ml/kg of clear fluid by mouth at 2-hour period before surgical scheduled time
  Interventions: Other: Clear oral fluid
- 5 ml/kg of clear oral fluid (Active Comparator): This group of patient will consume 5 ml/kg of clear fluid by mouth at 2-hour period before surgical scheduled time
  Interventions: Other: Clear oral fluid
- 7 ml/kg of clear oral fluid (Active Comparator): This group of patient will consume 7 ml/kg of clear fluid by mouth at 2-hour period before surgical scheduled time
  Interventions: Other: Clear oral fluid
- 10 ml/kg of clear oral fluid (Active Comparator): This group of patient will consume 10 ml/kg of clear fluid by mouth at 2-hour period before surgical scheduled time
  Interventions: Other: Clear oral fluid

INTERVENTIONS:
Other: Clear oral fluid — clear oral fluid including water, pulp-free juice and tea or coffee without milk.

SUMMARY:
According to the American Society of Anesthesiologists (ASA) fasting guideline for patients undergoing elective surgery, the 2-hour fasting period is suggested for clear oral fluid (including water, pulp-free juice and tea or coffee without milk). This guideline does not give any suggestions for proper volume of clear oral fluid intake.

This study is a prospective randomized control trials in children aged 13 through 17 years who are scheduled for an elective upper GI endoscopy procedure in the Gastroenteral Procedure Unit (GPU) at Boston Children's Hospital. The participants will be randomly assigned into one of four groups: Group 1 will consume 3 ml/kg of clear fluid by mouth at 2-hour period before surgical scheduled time, Group 2 will consume 5 ml/kg, Group 3 will consume 7 ml/kg, and Group 4 will consume 10 ml/kg. The investigators plan to recruit 72 patients in each group and 288 patients for the whole study. Research team will collect patient's demographic data, vital signs, information about their EGD procedure. Then actual volume of the stomach content and acidity will be measured from the content that is suctioned from patient's stomach during upper GI endoscopy procedure.

The investigators believe that the information from this study will help establish a comprehensive NPO guideline.

DETAILED DESCRIPTION:
The ASA and ESA practice guidelines recommend a 2-hour fasting period for clear fluid (including water, pulp-free juice and tea or coffee without milk), a 4- hour fasting period for breast milk and a 6-hour fasting period for non-human milk and solid food to reduce risks of pulmonary aspiration. While the ESA guideline suggests 3 ml/kg of clear oral fluids intake as a start point, the ASA does not suggest the allowable amount of ingested fluids/food volume.

According to the current consensus statement from the Association of Paediatric Anaesthetists of Great Britain and Ireland, the European Society of Paediatric Anaesthesiology and L'Association Des Anesthésistes-Réanimateurs Pédiatriques d'Expression Française on clear fluids fasting for elective pediatric general anesthesia in February 2018, this 3 ml/kg volume would mean patients ages 1-5 years old are allowed up to 55 ml, 6-12 years old up to 140 ml and greater than 12 years old up to 250 ml. The European consensus also suggests 1 hour clear fluid fasting for children as a practical way to reduce fasting times without increase aspiration risks.

To prevent preoperative dehydrated states which result in preoperative irritable behavior and intraoperative hypotension, patient fasting states and volume status should be optimized. Schmitz et al showed results of gastric emptying time of less than 30 minutes in healthy 6-14 years old children who had serial MRI scan every 30 minutes up to 120 minutes after drinking 7ml/kg of diluted raspberry syrup in 2011, the published clinical evidence suggested that clear fluids are absorbed to gastric volume of 1 ml/kg after 1 hour without pulmonary aspiration. Gawecka et al. also found no aspiration in ASA I and II children who were assigned to received 10ml/kg of 12.6% oral carbohydrate solution two hours before induction of anesthesia. Those studies showed no pulmonary aspiration event. However; pulmonary aspiration of gastric content is still a mainly concern for anesthesiologists when patients ingested large fluid volume. Previous studies reported incidences of aspiration range from1 to 10:10,000 cases and few cases require intensive care and respiratory support. The liberal clear fluid intake volume has been demonstrated to have similar risk of pulmonary aspiration as fasting patients.

The investigators propose a prospective randomized study on the relationship between assigned amount of clear oral fluid intake (ml/kg) and actual intra-gastric volume and pH of pediatric surgical patients. This study will be done at BCH's Gastroenterology Procedure Unit (GPU). Patients' demographic data will be obtained from charts. Patients will be randomly assigned to drink specific amount of fluid at 2 hours period before scheduled time. Patients or parents will be asked for other type, volume and time of last fluid/food intake. Actual intragastric volume and pH will be measured by the research team from the intragastric content that is removed at the beginning EGD procedures.

The investigators hope to demonstrate the relationship between volume of clear fluid intake at the 2-hour period before induction of anesthesia and actual intragastric volume which provide sufficient evidence of allowable clear fluid intake volume. Finally, the investigators want to use this study information to optimize standard fasting guidelines, to improve patients' preoperative volume status, to increase patient satisfaction and maintain patient safety.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification: I and II
* 13-17 years
* IPD cases or the first OPD case
* Scheduled for elective EGD procedure.
* All participants, families or guardians will be fluent in English.

Exclusion Criteria:

* Emergent EGD procedures
* Patients with active upper GI bleeding
* Patients who received preoperative oral medication
* Patients who are diagnosed as GERD, achalasia or suspected to have gastroparesis status such as uncontrolled diabetes or end stage kidney disease.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 288 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Gastric volume | We will collect data on a day of surgery from patient's arrival until they are discharged from PACU upto 24 hours
  Actual gastric content volume (ml) suctioned out of each pediatric patient's stomach

SECONDARY OUTCOMES:
Gastric pH | We will collect data on a day of surgery from patient's arrival until they are discharged from PACU upto 24 hours
  Actual gastric acidity (pH) suctioned out of each pediatric patient's stomach
Incidence of pulmonary aspiration | We will collect data on a day of surgery from patient's arrival until they are discharged from PACU upto 24 hours
  Pulmonary aspiration is defined by the presence of gastric contents in oral cavity or aspiration of gastric content into the larynx. This may cause a syndrome of progressive dyspnea, hypoxia, bronchial wheeze and patchy collapse and consolidation on chest X-ray.

CONTACTS AND LOCATIONS:
Overall Officials: Patcharee Sriswasdi, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
We might share IPD if it could maximize patient's benefit.

REFERENCES:
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Background] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Background] Maltby JR, Sutherland AD, Sale JP, Shaffer EA. Preoperative oral fluids: is a five-hour fast justified prior to elective surgery? Anesth Analg. 1986 Nov;65(11):1112-6. PMID 3767008
- [Background] Andersson H, Zaren B, Frykholm P. Low incidence of pulmonary aspiration in children allowed intake of clear fluids until called to the operating suite. Paediatr Anaesth. 2015 Aug;25(8):770-777. doi: 10.1111/pan.12667. Epub 2015 May 4. PMID 25940831
- [Background] Phillips S, Daborn AK, Hatch DJ. Preoperative fasting for paediatric anaesthesia. Br J Anaesth. 1994 Oct;73(4):529-36. doi: 10.1093/bja/73.4.529. PMID 7999497
- [Background] Dennhardt N, Beck C, Huber D, Sander B, Boehne M, Boethig D, Leffler A, Sumpelmann R. Optimized preoperative fasting times decrease ketone body concentration and stabilize mean arterial blood pressure during induction of anesthesia in children younger than 36 months: a prospective observational cohort study. Paediatr Anaesth. 2016 Aug;26(8):838-43. doi: 10.1111/pan.12943. Epub 2016 Jun 13. PMID 27291355
- [Background] Schmitz A, Kellenberger CJ, Liamlahi R, Studhalter M, Weiss M. Gastric emptying after overnight fasting and clear fluid intake: a prospective investigation using serial magnetic resonance imaging in healthy children. Br J Anaesth. 2011 Sep;107(3):425-9. doi: 10.1093/bja/aer167. Epub 2011 Jun 14. PMID 21676893
- [Background] Gawecka A, Mierzewska-Schmidt M. Tolerance of, and metabolic effects of, preoperative oral carbohydrate administration in children - a preliminary report. Anaesthesiol Intensive Ther. 2014 Apr-Jun;46(2):61-4. doi: 10.5603/AIT.2014.0013. PMID 24858963